CLINICAL TRIAL: NCT00494377
Title: Duloxetine Versus Duloxetine Plus Non-Pharmacological Intervention in the Treatment of Depression
Brief Title: Duloxetine Versus Duloxetine Plus Non-Drug Therapy for Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8601; F1J-MC-HMDD
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2007-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: duloxetine

SUMMARY:
The primary purpose of this study is to determine if duloxetine plus non-drug intervention is more effective than duloxetine alone in patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age who, in the opinion of the investigator, meet criteria for major depressive disorder (MDD) as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria.

Exclusion Criteria:

* Have a previous diagnosis of bipolar disorder, schizophrenia, or other psychotic disorders.
* Serious medical illness or clinically significant laboratory abnormalities that, in the judgment of the investigator, are likely to require medication/ intervention/hospitalization during the course of the study.
* Abnormal thyroid stimulating hormone (TSH) concentration (outside the reference range of the performing laboratory). Note: Patients diagnosed with hyperthyroidism or hypothyroidism who have been treated on a stable dose of thyroid supplement for at least the past 3 months, have medically appropriate TSH concentration, and are clinically euthyroid are allowed.
* Moderate or severe hepatic impairment, including but not limited to acute liver injury (such as hepatitis), and severe (Child-Pugh Class C) cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940
Dates: Start 2004-02; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To test whether duloxetine 60-120 mg daily, when combined with non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by remission rate (proportion of patients with HAMD17 score < or = 7 at endpoint)

SECONDARY OUTCOMES:
To test whether duloxetine 60-120 mg daily, when combined with non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone as measured by: Mean change (baseline to endpoint) on HAMD17
To test whether duloxetine 60-120 mg daily, when combined with non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by response rates (> or = 50% decrease from baseline to endpoint on HAMD17)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by HAMD17 subscales (Core, Maier, Anxiety/Somatization, Retardation/Somatization, Sleep & General Somatic Symptoms item)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by mean change from baseline to endpoint on the revised Mood and Physical symptoms of Depression scale (MAP-D)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by treatment adherence as measured by the Morisky Medication Adherence Questionnaire and study drug compliance
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Clinical Global Impression of Severity (CGI - Severity) Rating Scale
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Patient Global Impression of Improvement (PGI - Improvement) Rating Scale
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by patient satisfaction with medication and treatment overall as measured by a Visual Analogue Scale (VAS)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by attitudes to taking medicines as measured by the Beliefs about Medicines Questionnaire (BMQ)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Quality of Life and Health Outcome measure: EuroQol Questionnaire (EQ-5D)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Quality of Life and Health Outcome measure: Symptom Questionnaire
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Quality of Life and Health Outcome measure: Somatic Subscale (SQ-SS)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Quality of Life and Health Outcome measure: 36-item Short-Form Health Survey (SF-36)
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by Quality of Life and Health Outcome measure: Resource Use and Hospitalization Module
To test if duloxetine 60-120 mg daily + non-pharmacological intervention, is superior to duloxetine 60-120 mg daily alone, measured by painful physical symptoms of depression as measured by the VAS for Pain
To evaluate safety and tolerability of duloxetine 60-120 mg daily when combined with non-pharmacological intervention and duloxetine 60-120 mg daily alone, as measured by spontaneously reported treatment-emergent adverse events (TEAEs)
To evaluate the incidence of adverse events during Study Period III (optional taper period) as measured by spontaneously reported adverse events
To validate a revised version of the MAP-D (a novel scale for the measurement of emotional and physical symptoms of depression) in European outpatients with depression

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com